CLINICAL TRIAL: NCT04887974
Title: Canine Retraction Using Power Arms and Temporary Anchorage Devices
Brief Title: Canine Retraction With Temporary Anchorage Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Yehya Mostafa, Head of the Orthodontic Department, Future University in Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20153110
Record Dates: First submitted 2021-05-07; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Class II Malocclusion; Class III Malocclusion; Crowding, Tooth; Bimaxillary Protrusion
MeSH Terms: conditions — Overbite; Malocclusion, Angle Class III; Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Canine retraction (Experimental): The canines will be retracted by extending short silver elastomeric chains between the power arms in the canine brackets and the TADs. The applied force will be checked and adjusted to 150 g.
  Interventions: Procedure: canine retraction

INTERVENTIONS:
Procedure: canine retraction — Canine retraction using elastomeric chains activated every 4 weeks, using power arms to direct force through the center of resistance and TADs for direct anchorage.

SUMMARY:
Various malocclusions require the extraction of the first premolars and retraction of the canines with the need for maximum anchorage. If the canines are pulled into the extraction space using the molar teeth for support, unwanted tooth movement occurs. This study aims to evaluate the effect of temporary anchorage devices and power arms, which are auxiliary orthodontic appliances in reducing undesirable tooth movements.

DETAILED DESCRIPTION:
In orthodontic patients who require overjet correction, increased facial convexity, or relief of severe crowding, dental extraction followed by canine retraction is indicated. In conventional orthodontic treatment, the molars are used for anchorage and reinforced with intra-oral or extra-oral appliances. Although effective, this produces unwanted side effects where the molars move mesially and rotate, taking up some of the extraction space. As the canines move into the extraction space they tip backward requiring further uprighting. Power arms are vertical metal extensions placed in the canine brackets. They direct the force to the center of resistance of the tooth to allow bodily movement and prevent canine tipping. Temporary anchorage devices (TADs) are minimally invasive, small screws, inserted in the jaw bones to act as anchorage units instead of the molars.

This study aims to evaluate the effect of the TADs and power arms on the efficiency of canine retraction including the rate of canine retraction and canine tipping as well as mesial molar drift and rotation.

The null hypothesis is that the use of the power arm and the TADs have no effect on the canine retraction rate.

This study is a single-arm, single-center study. Twenty quadrants in 10 adult patients will be selected from the Orthodontic Outpatient Clinic at the Future University in Egypt.

Orthodontic records will be collected including study models, intra- and extra-oral photographs and cone beam computed tomograms.

Molars will be banded and Roth 0.22" brackets will be bonded to the canine and second premolars. Power arms, 8mmin length, will be inserted in the vertical slots of the canine brackets.

The dental arches will be leveled and aligned using consecutive archwires. TADs will be inserted between the second premolars and first molars. The first premolars will then be extracted and canines will be retracted within a week. Canines will be retracted along 0.016" X 0.22" stainless steel archwires using 150 g of force applied by an elastomeric chain. The elastic chain will be replaced every 4 weeks.

After 6 months of canine retraction, the orthodontic records will be collected for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Adult orthodontic patient
* Any malocclusion requiring the extraction of the first premolar and canine retraction
* Full permanent dentition with the exception of the wisdom teeth.

Exclusion Criteria:

* Any missing permanent tooth
* Previous orthodontic treatment
* Periodontal disease; pregnancy
* Systemic disease or medication that affects bone metabolism

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04-02 (Actual); Primary Completion 2017-01-14 (Actual); Study Completion 2017-01-14 (Actual)

PRIMARY OUTCOMES:
Canine retraction | Baseline to 6 months
  Amount of canine movement in millimeters measured on digital models. . The change in the vertical distance from the canine cusp tip to a line connecting the medial points of the third palatal rugae
Molar mesial drift | Baseline to 6 months
  Amount of molar movement in millimeters measured on digital models. The change in the vertical distance from the mesiobuccal cusp tip to a line connecting the medial points of the third palatal rugae

SECONDARY OUTCOMES:
Canine tipping | Baseline to 6 months
  The change in the angle between the canine long axis, from cusp tip to root apex, and the palatal plane (a plane passing through the incisive foramen and the anterior and posterior nasal spines); measued on the cone beam computed tomogram.
molar rotation | Baseline to 6 months
  The change in the angle between the molar horizontal axis and frontal Plane on the cone beam computed tomogram, in the axial view.

CONTACTS AND LOCATIONS:
Overall Officials: Yehya Mostafa, Study Director — Future University in Egypt
Locations (1):
- Faculty of Oral & Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No